CLINICAL TRIAL: NCT01533207
Title: A Phase III Randomized Trial of Gemcitabine (NSC# 613327) Plus Docetaxel (NSC# 628503) Followed by Doxorubicin (NSC# 123127) Versus Observation for Uterus-Limited, High Grade Uterine Leiomyosarcoma
Brief Title: Gemcitabine Hydrochloride and Docetaxel Followed by Doxorubicin Hydrochloride or Observation in Treating Patients With High-Risk Uterine Leiomyosarcoma Previously Removed by Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0277; NCI-2012-00249 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000724874; IRCI 001; GOG-0277; GOG-0277 (Other: NRG Oncology); GOG-0277 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2012-02-11; First posted 2012-02-15 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Stage I Uterine Sarcoma AJCC v7; Uterine Corpus Leiomyosarcoma
MeSH Terms: interventions — Watchful Waiting; Observation; Docetaxel; Doxorubicin; Filgrastim; Granulocyte Colony-Stimulating Factor; Gemcitabine; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (chemotherapy) (Experimental): Patients receive adjuvant gemcitabine hydrochloride IV over 70-90 minutes on days 1 and 8 and docetaxel IV over 30-60 minutes on day 8. Patients also receive filgrastim SC on days 9-15 or pegfilgrastim SC on day 9 or 10. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo CT and/or MRI. Patients with no evidence of disease receive doxorubicin hydrochloride IV every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive filgrastim SC on days 2-8 or pegfilgrastim SC on day 2 or 3.
  Interventions: Drug: Docetaxel; Drug: Doxorubicin Hydrochloride; Biological: Filgrastim; Drug: Gemcitabine Hydrochloride; Biological: Pegfilgrastim
- Arm II (no treatment) (Other): Patients undergo clinical observation.
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — Patients followed clinically
  Other Names: observation
  Arms: Arm II (no treatment)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm I (chemotherapy)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Arm I (chemotherapy)
Biological: Filgrastim — Given subcutaneously (SC)
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
  Arms: Arm I (chemotherapy)
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011
  Arms: Arm I (chemotherapy)
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Pegfilgrastim Biosimilar HSP-130; SD-01; SD-01 sustained duration G-CSF
  Arms: Arm I (chemotherapy)

SUMMARY:
This randomized phase III trial studies how well gemcitabine hydrochloride and docetaxel followed by doxorubicin hydrochloride work compared to observation in treating patients with high-risk uterine leiomyosarcoma previously removed by surgery. Drugs used in chemotherapy, such as gemcitabine hydrochloride, docetaxel, and doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether combination therapy after surgery is an effective treatment for uterine leiomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether overall survival of patients with uterus-limited high-grade leiomyosarcoma is superior among patients assigned to treatment with adjuvant gemcitabine hydrochloride (gemcitabine) plus docetaxel followed by doxorubicin hydrochloride compared to patients assigned to observation.

SECONDARY OBJECTIVES:

I. To determine whether treatment with adjuvant gemcitabine plus docetaxel followed by doxorubicin improves recurrence-free survival of patients with uterus-limited high-grade leiomyosarcoma compared to observation.

II. To explore the impact of potential predictors of recurrence or death such as patient age, institution reported tumor size, cervix involvement (yes or no), and mitotic rate.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive adjuvant gemcitabine hydrochloride IV over 70-90 minutes on days 1 and 8 and docetaxel IV over 30-60 minutes on day 8. Patients also receive filgrastim subcutaneously (SC) on days 9-15 or pegfilgrastim SC on day 9 or 10. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo computed tomography (CT) and/or magnetic resonance imaging (MRI). Patients with no evidence of disease receive doxorubicin hydrochloride IV every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive filgrastim SC on days 2-8 or pegfilgrastim SC on day 2 or 3.

Arm II: Patients undergo clinical observation.

After completion of study treatment, patients in both arms are followed up every 4 months for 3 years and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk uterine leiomyosarcoma (LMS), Federation of Gynecology and Obstetrics (FIGO) stage I (confined to corpus +/- cervix); patients with known uterine serosa involvement are not eligible; patients should have had, at least, a complete hysterectomy (including removal of the cervix); bilateral salpingo-oophorectomy is not required

  * Institutional pathology review calls the uterine leiomyosarcoma ?high grade?
  * Additionally, if the pathology report indicates a mitotic rate, the mitotic rate should be greater than or equal to 5 mitoses/10 high-power field
  * All patients must be no longer than 12 weeks (3 months) from surgical resection of cancer at the time of enrollment on study; if a patient requires a second operation to complete her surgery, i.e., trachelectomy to remove the cervix and/or bilateral salpingo-oophorectomy (BSO), the 12 weeks may be counted from the time of the second operation
  * Patients who had a ?morcellation? hysterectomy procedure that involved morcellation within the peritoneal cavity are eligible IF a second operation is performed and biopsies from the second procedure show no evidence of leiomyosarcoma
* All patients must have no evidence of persistent or metastatic disease as documented by a post-resection computed tomography (CT) of the chest/abdomen/pelvis or by CT chest + magnetic resonance imaging (MRI) abdomen/pelvis; the post-resection imaging studies should be performed within 4 weeks of registration on study
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcL (ANC >= 1.5 x 10^9/liter [L])
* Platelets greater than or equal to 100,000/mcL (platelets >= 100 x 10^9/L)
* Hemoglobin greater than 8.0 g/dL (= 80 g/L or 4.9 mmol/L)
* Creatinine less than or equal to 1.5 x institutional upper limit of normal (ULN)
* Bilirubin* within normal range
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST])* and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT])* less than or equal to 2.5 times ULN
* Alkaline phosphatase* less than or equal to 2.5 x ULN
* * Patients with a history of Gilbert?s syndrome may be eligible provided total bilirubin is less than or equal to 1.5 x ULN and the AST, ALT, and alkaline phosphatase meet the criteria detailed
* Neuropathy (sensory and motor) less than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Patients with Gynecologic Oncology Group (GOG) performance status of 0 or 1 OR Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1 OR Karnofsky performance status (PS) >= 80%
* Patients who have met the pre-entry requirements specified
* Patients must have signed an approved informed consent
* Patients participating through United States (U.S.) sites must sign an approved and authorization permitting release of personal health information
* Patients should be free of active infection requiring antibiotics (with the exception of an uncomplicated urinary tract infection [UTI])

Exclusion Criteria:

* Patients who have had prior therapy with docetaxel, gemcitabine hydrochloride, or doxorubicin hydrochloride at any time in their history
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are ineligible if there is any evidence of other malignancy being present within the last five years; patients are also ineligible if their previous cancer treatment contraindicates this protocol therapy
* Patients with a history of severe hypersensitivity reaction to Taxotere (docetaxel) or other drugs formulated with polysorbate 80
* Patients with GOG performance status of 2, 3 or 4; or ECOG performance status of 2, 3 or 4
* Patients who are breast-feeding
* Patients with a known history of congestive heart failure or cardiac ejection fraction < 50% (or less than institutional normal limits); echocardiogram (ECHO) or multigated acquisition scan (MUGA) is not required prior to enrollment; for patients assigned to the chemotherapy arm, an ECHO or MUGA should be done within 6 months of day 1 of gemcitabine-docetaxel treatment

  * Patients who enroll on study and are randomized to Regimen I (chemotherapy ) and then are found on baseline ECHO or MUGA to have cardiac ejection fraction < 50% or below institutional normal will remain ON study; such patients will receive gemcitabine + docetaxel for 4 cycles but will NOT receive any doxorubicin treatment; they will continue treatment follow-up as outlined for all patients assigned to Regimen I
* Patients with a history of prior whole pelvic radiation
* Concurrent treatment with hormone replacement therapy is permitted at the discretion of the treating physician; patients who have been taking hormonal/hormone blocking agents for breast cancer or breast cancer prevention or other indication are eligible; use of anti-hormonal agents (tamoxifen, medroxyprogesterone, aromatase inhibitors) is permitted at the discretion of the treating physician; documentation of concurrent medications is required
* Patients with recurrent uterine LMS
* Patients who are known to be human immunodeficiency virus (HIV) positive are not eligible
* Patients with gross residual or metastatic tumor findings following complete surgical treatment for uterine LMS

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martee L Hensley, Principal Investigator — NRG Oncology
Locations (623):
- United States (608):
  - Tennessee Valley Gynecologic Oncology, Huntsville, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute Altamonte, Altamonte Springs, Florida
  - Florida Hospital Kissimmee, Kissimmee, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Florida Urology Associates-Orlando, Orlando, Florida
  - Florida Hospital East Orlando, Orlando, Florida
  - Florida Hospital Cancer Institute Winter Park, Winter Park, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Randolph Hospital, Asheboro, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Matthews Radiation Oncology Center, Matthews, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Virginia Mason Bainbridge Island Medical Center, Bainbridge Island, Washington
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Virginia Mason Federal Way Medical Center, Federal Way, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Tacoma/Valley Radiation Oncology Centers-Gig Harbor, Gig Harbor, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Northwest Cancer Clinic, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Virginia Mason Lynnwood Medical Center, Lynnwood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Peninsula Cancer Center, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Tacoma/Valley Radiation Oncology Centers-Puyallup, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - Tacoma/Valley Radiation Oncology Centers-Jackson Hall, Tacoma, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Tacoma/Valley Radiation Oncology Centers-Saint Joe's, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Monongalia Hospital, Morgantown, West Virginia
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- France (4):
  - Institut Bergonie Cancer Center, Bordeaux
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Centre Catherine de Sienne, Nantes
- University Medical Center Groningen, Groningen, Netherlands
- University of Oslo, Oslo, Norway
- Hospital Clinico San Carlos, Madrid, Spain
- United Kingdom (6):
  - Addenbrookes Hospital-Medical School, Cambridge, England
  - University College London Hospital, London, England
  - Christie Hospital, Manchester, England
  - Weston Park Hospital, Sheffield, England
  - Beatson Oncology Center, Glasgow, Scotland
  - Institute of Cancer Research - Chelsea, London
- Hospital Universitario, Caracas, Venezuela

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study accrued 38 patients from June 2012 to September, 2016. Study was closed due to accrual futility.
Groups:
- Regimen 1: Gemcitabine 900 mg/m2 IV days 1 and 8 Docetaxel 75 mg/m2 IV day 8 GCSF 5 micrograms/kg days 9-15 or pegfilgrastim 6 mg day 9 or 10 Every 21 days for 4 cycles CT/MRI imaging to confirm disease-free Doxorubicin 60 mg/m2 IV every 21 days for 4 cycles
- Regimen II: Observation
Period: Overall Study
Arm/Group | Regimen 1 | Regimen II
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Regimen II | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 0 | 0 | 0
  30-39 years | 2 | 0 | 2
  40-49 years | 4 | 4 | 8
  50-59 years | 10 | 7 | 17
  60-69 years | 3 | 5 | 8
  70-79 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 15 | 11 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Death
Description: The duration of time from study entry to time of death or the date of last contact.
Time Frame: Follow-up every 4 months for 3 years, then every 6 months for 2 years.
Population: Eligible and evaluable participants
Measure: Number; unit: Participants
Arm/Group | Regimen 1 | Regimen II
Number analyzed (Participants) | 20 | 18
Participants | 5 | 1

2. Secondary Outcome: Incidence of Grade 3 or Higher Adverse Events as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Time Frame: Approximately 4 years
Population: eligible and randomized patients
Measure: Number; unit: participants
Arm/Group | Regimen 1 | Regimen II
Number analyzed (Participants) | 20 | 18
participants | 10 | 1

3. Secondary Outcome: Number of Participants With Recurrence
Description: The duration of time from study entry to time of recurrence or death, whichever occurred first, or the date of last contact.
Time Frame: Follow-up every 4 months for 3 years, then every 6 months for 2 years.
Population: Eligible and evaluable participants
Measure: Number; unit: participants
Arm/Group | Regimen 1 | Regimen II
Number analyzed (Participants) | 20 | 18
participants | 8 | 8

4. Other Pre Specified Outcome: Univariate and Multi-variable Prognostic Significance of Baseline Clinical, Pathologic, or Demographic Factors
Description: Analyses will be carried out using proportional hazards models of both survival and recurrence.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For Regimen 1: Baseline (pre-treatment); Prior to each cycle of chemotherapy, up to 4 months. For Regimen 2: Every 3-4 weeks for months 1-3. Every 3-4 weeks for months 3-6 on study.
Arm/Group | Regimen 1 | Regimen II
All-Cause Mortality (participants affected / at risk) | 5/20 | 1/18
Serious Adverse Events (participants affected / at risk) | 5/20 | 0/18
Other Adverse Events (participants affected / at risk) | 16/20 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (N=20) | Regimen II (N=18)
Mucositis Oral (Gastrointestinal disorders) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Catheter Related Infection (Infections and infestations) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (N=20) | Regimen II (N=18)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 3 | 0
Anemia (Blood and lymphatic system disorders) | 13 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 4 | 1
Chest Pain - Cardiac (Cardiac disorders) | 1 | 0
Hearing Impaired (Ear and labyrinth disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Watering Eyes (Eye disorders) | 2 | 0
Blurred Vision (Eye disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 6 | 1
Diarrhea (Gastrointestinal disorders) | 7 | 1
Vomiting (Gastrointestinal disorders) | 4 | 1
Bloating (Gastrointestinal disorders) | 2 | 1
Anal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 4 | 4
Mucositis Oral (Gastrointestinal disorders) | 5 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 12 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
General Disorders And Administration Site Conditio (General disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Malaise (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Edema Limbs (General disorders) | 7 | 2
Fatigue (General disorders) | 14 | 5
Fever (General disorders) | 6 | 0
Chills (General disorders) | 1 | 0
Infusion Related Reaction (General disorders) | 2 | 0
Infections And Infestations - Other (Infections and infestations) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 2 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 1 | 0
Phlebitis Infective (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Weight Gain (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 7 | 0
Creatinine Increased (Investigations) | 2 | 0
Neutrophil Count Decreased (Investigations) | 8 | 0
White Blood Cell Decreased (Investigations) | 7 | 0
Aspartate Aminotransferase Increased (Investigations) | 4 | 0
Alkaline Phosphatase Increased (Investigations) | 3 | 0
Alanine Aminotransferase Increased (Investigations) | 5 | 0
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Nervous System Disorders - Other (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 5 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 3
Dysgeusia (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 1
Akathisia (Nervous system disorders) | 1 | 0
Personality Change (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Depression (Psychiatric disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 3 | 3
Urine Discoloration (Renal and urinary disorders) | 1 | 0
Urinary Urgency (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 2 | 1
Urinary Tract Pain (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal Inflammation (Reproductive system and breast disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 11 | 1
Surgical And Medical Procedures - Other (Surgical and medical procedures) | 1 | 0
Thromboembolic Event (Vascular disorders) | 3 | 0
Superficial Thrombophlebitis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 2
Hot Flashes (Vascular disorders) | 4 | 4
Flushing (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was closed early due to slow participant accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT01533207/Prot_SAP_000.pdf